CLINICAL TRIAL: NCT04853030
Title: A Double-blind, Multinational, Multicentre, Randomised, 2-period Crossover Study to Assess the Efficacy and Safety of Advanced Closed-loop Insulin Delivery With Minimed 670 4.0 System Comparing Faster Insulin Aspart to Standard Insulin Aspart Therapy Over 4 Weeks in Active Children and Adolescents With Type 1 Diabetes - the FACT Study
Brief Title: Fast Advanced Closed-Loop Therapy
Acronym: FACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Collaborators: Medical University of Graz Department of Pediatrics and Adolescent Medicine, Graz, Austria (Unknown); UMC Ljubljana University Children's Hospital Ljubljana (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FACT Study
Record Dates: First submitted 2021-04-07; First posted 2021-04-21 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded insulin formulation (Faster and Standard Insulin Aspart)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimed 670G 4.0 closed loop with Faster Insulin aspart (Experimental)
  Interventions: Drug: Fiasp
- Minimed 670G 4.0 closed loop with Standard Insulin aspart (Active Comparator)
  Interventions: Drug: Novorapid

INTERVENTIONS:
Drug: Fiasp — Advanced closed-loop insulin therapy with Faster acting insulin Aspart (Fiasp)
  Arms: Minimed 670G 4.0 closed loop with Faster Insulin aspart
Drug: Novorapid — Advanced closed-loop insulin therapy with Standard acting insulin Aspart (Novorapid
  Arms: Minimed 670G 4.0 closed loop with Standard Insulin aspart

SUMMARY:
A double-blind, multinational, multicenter, randomised, 2-period crossover study to assess the efficacy and safety of advanced closed-loop insulin delivery with Minimed 670G 4.0 system comparing Faster Insulin Aspart to Standard Insulin Aspart therapy over 4 weeks in active children and adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 and 18 years of age
* Type 1 diabetes for at least 6 months
* Insulin pump user for at least 3 months
* Total daily dose of insulin >8 units/day
* Treated with rapid acting insulin analogue
* Subject/carer is willing to perform at least 2 finger-prick blood glucose measurements per day
* Screening HbA1c ≤ 11 % (97 mmol/mol) based on analysis from local laboratory
* Willing to wear glucose sensor
* Willing to wear closed loop system 24/7
* The subject is willing to follow study specific instructions
* The subject/carer is willing to upload pump and CGM data at regular intervals

Exclusion Criteria:

* Physical or psychological disease likely to interfere with normal conduct of the study
* Untreated coeliac disease or thyroid disease
* Current treatment with drugs known to interfere with glucose metabolism
* Participation in another interventional clinical investigation
* Treated with ultra-rapid acting insulin analogue
* Known or suspected allergy to insulin
* Carer's lack of reliable telephone facility for contact
* Subject's severe visual impairment
* Subject's severe hearing impairment
* Medically documented allergy towards the adhesive (glue) of plasters or subject is unable to tolerate tape adhesive in the area of sensor placement
* Serious skin diseases located at places of the body corresponding with sensor insertion sites
* Sickle cell disease, haemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Time above range 180 mg/dl | 12 weeks for each arm of the crossover
  The primary outcomes is a difference in CGM-measured metrics between periods (Minimed 670G 4.0 closed loop with Faster Insulin aspart and Minimed 670G 4.0 closed loop with Standard Insulin aspart) in superiority for proportion of time >180 mg/dL (10.0 mmol/L)

SECONDARY OUTCOMES:
Time in range 70-180 mg/dl | 4 weeks for each arm of the crossover
  CGM derived indices over the study period of each treatment period ((Minimed 670G 4.0 closed loop with Faster Insulin aspart and Minimed 670G 4.0 closed loop with Standard Insulin aspart)) for 24/7 in time in range 70 to 180 mg/dL (3.9 to 10.0 mmol/L
Time below range <70 mg/dl | 4 weeks for each arm of the crossover
  CGM derived indices over the study period of each treatment period ((Minimed 670G 4.0 closed loop with Faster Insulin aspart and Minimed 670G 4.0 closed loop with Standard Insulin aspart)) for 24/7 in time below range 70 mg/dl
Mean glucose | 4 weeks for each arm of the crossover
  CGM derived indices over the study period of each treatment period ((Minimed 670G 4.0 closed loop with Faster Insulin aspart and Minimed 670G 4.0 closed loop with Standard Insulin aspart)) for 24/7 in mean glucose

CONTACTS AND LOCATIONS:
Locations (2):
- Medical University of Graz Department of Pediatrics and Adolescent Medicine, Graz, Austria
- UMC Ljubljana University Children's Hospital Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dovc K, Bergford S, Frohlich-Reiterer E, Zaharieva DP, Potocnik N, Muller A, Lenarcic Z, Calhoun P, Fritsch M, Sourij H, Bratina N, Kollman C, Battelino T. A Comparison of Faster Insulin Aspart with Standard Insulin Aspart Using Hybrid Automated Insulin Delivery System in Active Children and Adolescents with Type 1 Diabetes: A Randomized Double-Blind Crossover Trial. Diabetes Technol Ther. 2023 Sep;25(9):612-621. doi: 10.1089/dia.2023.0178. PMID 37404205